CLINICAL TRIAL: NCT02389556
Title: Serum ANGPTL3, ANGPTL8 and Glypican 4 Concentrations in Relation to the Development of Obesity in Korean Children: a Three Year Prospective Cohort Study
Brief Title: Serum ANGPTL3, ANGPTL8 and Glypican 4 Concentrations in Relation to the Development of Obesity in Korean Children
Status: Completed | Type: Observational
Sponsor: Korea University (Other)
Responsible Party: Principal Investigator, Kyung Mook Choi, Professor of Endocrinology and Metabolism in Korea university, Korea University
Other Study IDs: KMOSES
Record Dates: First submitted 2015-03-10; First posted 2015-03-17 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples Without DNA — Serum was obtained from each subject after the subjects had fasted overnight for more than 8 hrs.
Oversight: Data Monitoring Committee: No

SUMMARY:
ANGPTL3 and ANGPTL8 are emerging molecules involving lipid metabolism. In previous in vivo study using mice, ANGPTL8 regulated the activation of ANGPTL3 which was known to inhibit lipoprotein lipase activity and stimulate lipolysis of adipose tissue. Besides, glypican 4 was identified as a novel adipokine modulating adipocyte differentiation. Thus, the investigators postulated that different serum concentrations of ANGPTL3, ANGPTL8 and glypican 4 might affect progression of obesity in children. The investigators measure these molecules in Korean children, and investigate the association between these molecules and development of obesity.

DETAILED DESCRIPTION:
Participants in this study were selected from the Korean Metabolic disorders & Obesity Study in Elementary School children (KMOSES), the main aim of which was to comprehensively assess obesity-related metabolic risk factors and to evaluate clinical outcomes in Korean children prospectively. Korean children who were participated in a school-based health examination, were reexamined for the 3-year follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were reexamined for the 3 year follow-up assessment

Exclusion Criteria:

* Participants who were not being available for the 3 year follow up assessment

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants in this study were selected from the Korean Metabolic disorders & Obesity Study in Elementary School children (KMOSES).
Sampling Method: Probability Sample
Enrollment: 457 (Actual)
Dates: Start 2006-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The changes of body mass index according to serum level of ANGPTL3, ANGPTL8 and glypican 4 | Baseline and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Kyung Mook Choi, MD, Principal Investigator — Department of Internal Medicine, Korea University College of Medicine
Locations (1):
- Department of Internal Medicine, Korea University College of Medicine, Seoul, VD, South Korea

IPD SHARING:
Plan to Share IPD: No